CLINICAL TRIAL: NCT04920136
Title: Gain of Keratinized Mucosa Around Teeth and Dental Implants Using a Combination of Strip Gingival Graft and Acellular Dermal Matrix
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hussein Basma, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300006910; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Gingival Recession; Lack of Keratinized Attached Peri-implant Mucosa; Thin Gingiva
Keywords: Attached mucosa; Keratinized tissue; Dental implants; Connective tissue
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strip Free gingival graft (SGG) + Acellular Dermal Matrix graft (ADM) (Experimental): A horizontal incision is then placed at the middle of residual KT. Two vertical releasing incisions are followed to allow for apical displacement of the flap. The recipient site should ideally retain intact periosteum that is firmly attached to bone with no loose fibers, no irregularities and no perforations.
  A strip of a free gingival graft is then harvested from the patient's palate. This strip is only 2 to 3 mm wide ,1 to 1.5 mm thick and has an appropriate length to cover the full apical extension of the recipient site. The strip is sutured immediately with 6-0 monocryl sutures. Coronal to the strip, the periosteal bed is covered with ADM, which is already rehydrated in sterile saline for 10 min, trimmed and customized to fit the available space. The ADM is then stabilized on the periosteal bed with the epithelium side facing upward. The ADM is fixed on the recipient bed by periosteal 6-0 monocryl sutures.
  Interventions: Procedure: Strip Free gingival graft (SGG) + Acellular Dermal Matrix graft (ADM)
- Free gingival graft. (Active Comparator): Two vertical incisions are made, and a partial thickness flap are designed to provide a firm and immobile periosteal bed. The raised partial thickness flap will be excised. Muscle and unattached connective tissue fibers are thoroughly scraped with a scalpel to prevent graft mobility. Autogenous FGG was harvested with #15C scalpel blade from hard palate at the same side randomly selected to receive the FGG. Donor area will be sutured with 5-0 gut sutures. FGG, is placed and stabilized with simple interrupted 5-0 vicryl sutures at recipient site coronal border and horizontal or periosteal anchorage sutures over the graft.
  Interventions: Procedure: Free Gingival graft

INTERVENTIONS:
Procedure: Strip Free gingival graft (SGG) + Acellular Dermal Matrix graft (ADM) — A horizontal incision is then placed at the middle of residual KT. Two vertical releasing incisions are followed to allow for apical displacement of the flap. The flap will be then elevated with a split-thickness flap beyond the mucogingival junction where it is sutured at this apical position using a mattress (5-0, monocryl) suture. The recipient site should ideally retain intact periosteum that is firmly attached to bone with no loose fibers, no irregularities and no perforations.
  Arms: Strip Free gingival graft (SGG) + Acellular Dermal Matrix graft (ADM)
Procedure: Free Gingival graft — Two vertical incisions are made, and a partial thickness flap are designed to provide a firm and immobile periosteal bed. The raised partial thickness flap will be excised. Muscle and unattached connective tissue fibers are thoroughly scraped with a scalpel to prevent graft mobility. Autogenous FGG was harvested with #15C scalpel blade from hard palate at the same side randomly selected to receive the FGG. Donor area was sutured with 5-0 gut sutures. FGG, is placed and stabilized with simple interrupted 5-0 vicryl sutures at recipient site coronal border and horizontal or periosteal anchorage sutures over the graft.
  Arms: Free gingival graft.

SUMMARY:
This study is to compare the two techniques to achieve change in the tissue quality at areas of lack of Keratinized Tissue (KT) using soft tissue grafting with autogenous graft material (Free Gingival Graft)(FGG) vs Strip gingival graft with acellular dermal matrix (ADM) (SGG+ADM).

DETAILED DESCRIPTION:
This investigation is a randomized controlled trial of two techniques to achieve change in the tissue quality at areas of lack of Keratinized Tissue (KT) using soft tissue grafting with autogenous graft material (Free Gingival Graft)(FGG) vs Strip gingival graft with acellular dermal matrix (ADM) (SGG+ADM). To evaluate to determine if either grafting technique (FGG vs SGG+ADM) demonstrates superiority in clinical (amount of KT increase, tissue thickness increase, and practitioner-assessed esthetics) and patient-centered outcomes (pain, swelling, change in daily activities, and patient-assessed esthetics) in a controlled study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Able to read and understand informed consent document
* Patients with teeth/implants lacking keratinized tissue.
* Must be a patient of the UAB Dental School
* Presence of periodontally healthy, non-carious neighboring teeth, healthy implants or edentulous ridges on either side of the involved site(s)

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Presence of active periodontal disease
* Previous soft tissue grafting at the site(s) to be treated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of soft tissue regenerated | From baseline to 12 months
  Compare the change in soft tissue quality (attached or keratinized ) between two used soft tissue grafts by superimposing the before and after intraoral scans and the calculating using a software the difference of soft tissue gain between both scans in (mm)
Quantity of soft tissue regenerated (Width of Keratinized Tissue) | From baseline to 12 months
  Using a periodontal probe , the width of keratinized tissue will be measured in (mm) and compared between two grafts used.

CONTACTS AND LOCATIONS:
Locations (1):
- Unversity of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No